CLINICAL TRIAL: NCT04041960
Title: Examining the Effects of Theta Burst Stimulation on the Neural Network Associated With Reading in Adult Struggling Readers
Brief Title: Effects of TBS on Reading in Adult Struggling Readers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgia State University (Other)
Collaborators: Medical University of South Carolina (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, C. Nikki Arrington, Principal Investigator, Georgia State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: H18271
Record Dates: First submitted 2019-07-29; First posted 2019-08-01 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: Developmental Reading Disorder; Dyslexia, Developmental
MeSH Terms: conditions — Dyslexia | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SMG (Experimental): Brain region targeted with transcranial magnetic stimulation: superamarginal gyrus
  Interventions: Other: Transcranial magnetic stimulation (TMS)
- MTG (Experimental): Brain region targeted with transcranial magnetic stimulation: middle temporal gyrus
  Interventions: Other: Transcranial magnetic stimulation (TMS)
- Vertex (Active Comparator): Brain region targeted with transcranial magnetic stimulation (none associated): Vertex
  Interventions: Other: Transcranial magnetic stimulation (TMS)

INTERVENTIONS:
Other: Transcranial magnetic stimulation (TMS) — The TMS protocol to be used, excitatory intermittent theta burst stimulation (iTBS), has been shown to have minimal risk in children as young as 6 (Hong et al., 2015), as well as adults (Huang et al., 2005). This stimulation paradigm uses a series of theta burst stimulation (TBS) units. Each unit consists of 3 pulses of stimulation given at 50 Hz (Huang et al., 2005). Excitatory iTBS consists of 20 sets of 10 TBS units (2 second duration) repeated every 10 seconds for a total of 190 seconds. One session of excitatory stimulation delivers a total of 600 pulses.

SUMMARY:
The purpose of this project is to understand how reading is related to brain function. To do this, participants will perform some reading tasks and then have magnetic resonance imaging (MRI) brain scans. Participants will then receive transcranial magnetic stimulation (TMS) to the reading areas of the brain, followed by a second MRI brain scan. This will temporarily activate reading abilities. We want to better understand how the reading system in the brain functions.

DETAILED DESCRIPTION:
Subjects will come in for up to 2 sessions, each lasting between 1 - 4 hours. Subjects will complete reading and cognitive tasks associated with reading, and receive TMS as well as 2 MRI brain scans, in order to assess brain regions important to reading.

Initial, basic screening including MRI and TMS safety screening will be conducted over the phone during the recruitment phone call and/or screening forms will be emailed to prospective subjects for their review. Those individuals that qualify will be scheduled for session 1. Session 1 will take between 1 and 3 hours. Subjects who pass health/MRI/TMS screening will complete cognitive/reading screening measures as well as the demographic information survey. They will also be trained on the MRI and TMS procedures. If all screening criteria is met, subjects will be asked to return for a second session which will include the MRI and TMS portions of the study.

Session 2 will take place on a separate day and consist of renewal of the health/MRI/TMS screening forms prior to the MRI scan or TMS administration. The baseline MRI portion of the session will last approximately 1.5 hours including screening, training, and scan time. The MRI scan will be followed by the TMS portion which will last approximately 45 minutes. The post-TMS MRI will take place immediately following the TMS session and will last approximately 45 minutes. Reading assessments will be administered before the baseline MRI and again after TMS stimulation/before post-TMS MRI, each lasting approximately 10 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Must meet the study reading criteria based on their reading and reading-related screening test results
* native speakers of English
* Right handed
* minimum of low average intellectual functioning (SS>=80) on at least one subscale on the Wechsler Abbreviated Scale of Intelligence-2

Exclusion Criteria:

* hearing deficits (>25dB at 500+ Hz), visual deficits (>20/40), serious emotional problems, certain neurological conditions (e.g., uncontrolled seizure disorders)
* Braces on teeth, a cardiac pacemaker; hearing aid; other metal in their body or eyes (which may include certain metallic-embedded tattoos), including but not limited to pins, screws, shrapnel, plates, dentures or other metal objects
* TMS or MRI Screening and Contraindication Forms which do not pass technician review

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Change in lexical decision making | 10 minutes after TMS
  Subjects will complete one computerized lexical decision making task before and after TMS stimulation in order to assess change in lexical decision making ability 10mins post stimulation. Subjects will see a word cue on the screen and asked to judge with a button press if the word cue is a "real word" or "not a real word."
Change in real-word reading efficiency | 5 minutes after TMS
  Subjects will complete a timed real word reading task before and after TMS stimulation in order to assess change in word reading ability 5mins post stimulation.; Subjects will read a list of words as quickly and as accurately as possible.
Change in Pseudoword reading efficiency | 5 to 10 minutes after TMS
  Subjects will complete a pseudoword reading task before and after TMS stimulation in order to assess change in pseudoword reading ability 5mins post stimulation. Subjects will read a list of pseudowords as quickly and as accurately as possible.
Change in phonemic decoding | 5 to 10 minutes after TMS
  Subjects will complete one computerized lexical phonemic decoding task before and after TMS stimulation in order to assess change in phonemic decoding ability 10mins post stimulation. Subjects will see a non-real word cue on the screen and be asked to judge with a button press if the non-real word cue can be pronounced like ("sounds like") a real word or not a real word.

SECONDARY OUTCOMES:
Change in function of neural reading network | 20 minutes after TMS
  Subjects will complete a functional MRI task requiring the subject to read a word and identify if it matches a picture present on the screen. This will be used to assess the effectiveness of the TMS on the targeted reading network.

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Advanced Brain Imaging, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD will be available via the Collaborative Informatics and Neuroimaging Suite data exchange
Supporting Information: Study Protocol, ICF
Time Frame: Data will be made available by January 2022 and will remain in COINS data exchange indefinitely.
Access Criteria: Request must be made via COINS data exchange
URL: https://coins.trendscenter.org/

REFERENCES:
- [Derived] Herrera-Diaz A, Bledniak E, Harrington RM, Morris R, Arrington CN. Functional Activation following Transcranial Magnetic Stimulation in Neurotypical Adult Readers. J Integr Neurosci. 2025 Mar 20;24(3):26365. doi: 10.31083/JIN26365. PMID 40152566